CLINICAL TRIAL: NCT03632551
Title: Localization and Mismatch Negativity in Subjects With Single-sided Deafness Ads Subjects With Unilateral Cochlear Implant
Brief Title: Localization and Mismatch Negativity
Acronym: MMNLocA
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University Hospital, Toulouse (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: RC31/18/0096
Record Dates: First submitted 2018-07-19; First posted 2018-08-15 (Actual); Last update posted 2023-08-23 (Actual); Status verified 2023-08

CONDITIONS: Deafness
Keywords: Mismatch negativity; EEG; Single sided deafness; Cochlear implant; Asymmetrical hearing loss; Spatial hearing; Binaural hearing; Localization
MeSH Terms: conditions — Deafness

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Symmetrical hearing (Active Comparator): Specific binaural hearing evaluations (recognition of sentences in noise, sound source localization) and quality of life (SSQ questionnaire) will be carried out. Thereafter, the electroencephalographic examination will be performed
  Interventions: Other: Specific binaural hearing evaluations
- Single-sided deafness (Experimental): Specific binaural hearing evaluations (recognition of sentences in noise, sound source localization) and quality of life (SSQ questionnaire) will be carried out. Thereafter, the electroencephalographic examination will be performed
  Interventions: Other: Specific binaural hearing evaluations
- Bilateral profound hearing loss treated (Experimental): Specific binaural hearing evaluations (recognition of sentences in noise, sound source localization) and quality of life (SSQ questionnaire) will be carried out. Thereafter, the electroencephalographic examination will be performed
  Interventions: Other: Specific binaural hearing evaluations

INTERVENTIONS:
Other: Specific binaural hearing evaluations — Specific binaural hearing evaluations (recognition of sentences in noise, sound source localization) and quality of life (SSQ questionnaire) will be carried out. Thereafter, the electroencephalographic examination will be performed

SUMMARY:
This descriptive and observational research project aims to characterize MMN as a neuronal marker of localization deficit in single-sided deafened subjects and subjects with bilateral profound deafness treated by a cochlear implant (CI). It includes several electro-physiological and psychoacoustic assessments performed on subjects with single-sided deafness and cochlear implanted subjects, with normal-hearing subjects as control:

* Evaluation of the characteristics of the MMN involved in sound localization by EEG.
* Evaluation of the spatial localization abilities for a sound source presented in the open field.
* Assessment of performance for speech recognition in noise. These evaluations are performed in subjects with symmetrical hearing, in a natural binaural condition and a monaural condition (with a plugged ear), in subjects with single-sided deafness and in subjects with unilateral CI

DETAILED DESCRIPTION:
Sound localization is the primary function of binaural hearing and facilitates speech recognition in noise. In case of unilateral or asymmetrical hearing loss, speech recognition in noise requires a constant adaptation of the head position to compensate for deafness. There is a significant impact of these deficits for socio-professional integration with a globally reduced quality of life . A researcher has found a significant correlation between performance for speech recognition in noise and the level of quality of life level assessed by a Spatial and Qualitative Hearing Scale (SSQ).

Subjects with bilateral profound deafness treated with cochlear implant (CI) usually recover excellent scores for speech recognition in quiet conditions. Nevertheless, hearing restoration is only partial and binaural hearing includes the fields where hearing remains impaired, as illustrated by the studies on sound localization or speech recognition in noise.

Studies using functional MRI, MEG or EEG to investigate neuro-functional reorganization following single-sided deafness show a reduced asymmetry in the hemispherical processing of auditory information, documented by an increase of cortical activity ipsilateral to the better ear, whether it is lateralized to right or left. However, the neural modifications underlying spatial hearing processing have hardly not been explored.

The mismatch negativity (MMN) is a specific potential, evoked by an auditory stimulation using two sounds almost similar. The presence of this MMN indicates that the auditory system is able to discriminate these 2 sounds, regardless of the subjective feedback reported by the subject.

The use of MMN to describe neural reorganization following cochlear implantation is expanding. Stimuli as diverse as pure sounds, tonal bursts or phonemes may be used, but to the investigator's knowledge there is no study investigating localization processes

ELIGIBILITY:
Inclusion Criteria:

For symmetrical hearing subjects:

* Affiliation to a social security
* Normal hearing, or mild to moderate symmetrical hearing loss controlled by tone audiometry performed before inclusion (in air conduction and bone conduction, frequencies 250 Hz to 4000 Hz).
* Signature of the consent form

For subjects with single-sided deafness:

* Affiliation to a social security
* Subject having a unilateral deafness controlled by pure-tone audiometry before inclusion (in air conduction and bone conduction, frequencies 250 Hz to 4000 Hz).
* Signature of the consent form

For subjects with Cochlear Implants:

* Affiliation to a social security
* Subject with symmetrical or asymmetrical profound deafness treated by unilateral cochlear implantation.
* Signature of the consent form

Exclusion Criteria:

* History of associated neurological disorder
* Taking psychotropic drugs
* Persons with complicated social or medical situations

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2018-07-10 (Actual); Primary Completion 2020-12-10 (Actual); Study Completion 2023-12 (Estimated)

PRIMARY OUTCOMES:
Characterization of the MMN in the group of subjects with single-sided deafness and the group of CI subjects | Inclusion visit
  Amplitude and latency in MMN recordings

SECONDARY OUTCOMES:
Performances for sound source localization and speech recognition in noise across the different groups | Inclusion visit
  Critical signal-to-noise ratios (SRT for speech reception threshold, signal-to-noise ratio authorizing the correct discrimination of 50 % of the words) obtained in the test of discrimination of the word in the presence of a rival noise MATRIX in condition dichotique, diotique and dichotique inverted.
Speech Spatial Quality of the subjects according to the study group | Inclusion visit
  Speech Spatial Quality (SSQ) questionnaire
Correlation between the characteristics of the localization MMN, the behavioral performances for sound source localization and the speech recognition in noise, and the level of quality of life according to the study group | Inclusion visit
  Coefficient of correlation between the characteristics of the MMN of location and the performances of location Coefficient of correlation between the characteristics of the MMN of location and the SRT obtained in the test of discrimination of the word Coefficient of correlation between the characteristics of the MMN of location and the score obtained in the SSQ

CONTACTS AND LOCATIONS:
Overall Officials: Mathieu Marx, PU-PH, Principal Investigator — University Hospital, Toulouse
Locations (1):
- Oto rhino laryngologie, Toulouse, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Avan P, Giraudet F, Buki B. Importance of binaural hearing. Audiol Neurootol. 2015;20 Suppl 1:3-6. doi: 10.1159/000380741. Epub 2015 May 19. PMID 25998698
- [Background] Baguley DM, Humphriss RL, Axon PR, Moffat DA. The clinical characteristics of tinnitus in patients with vestibular schwannoma. Skull Base. 2006 May;16(2):49-58. doi: 10.1055/s-2005-926216. PMID 17077869
- [Background] Bennemann J, Freigang C, Schroger E, Rubsamen R, Richter N. Resolution of lateral acoustic space assessed by electroencephalography and psychoacoustics. Front Psychol. 2013 Jun 11;4:338. doi: 10.3389/fpsyg.2013.00338. eCollection 2013. PMID 23781211
- [Background] Budinger E, Brechmann A, Brosch M, Heil P, Konig R, Ohl FW, Scheich H. Auditory cortex 2014 - towards a synthesis of human and animal research. Eur J Neurosci. 2015 Mar;41(5):515-7. doi: 10.1111/ejn.12832. No abstract available. PMID 25728172
- [Background] Chan JC, Freed DJ, Vermiglio AJ, Soli SD. Evaluation of binaural functions in bilateral cochlear implant users. Int J Audiol. 2008 Jun;47(6):296-310. doi: 10.1080/14992020802075407. PMID 18569102